CLINICAL TRIAL: NCT03782324
Title: Mechanical Complications After Central Venous Catheterisation
Acronym: CVC-MECH
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: CVC-MECH
Record Dates: First submitted 2018-12-04; First posted 2018-12-20 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Mechanical Complications of Central Venous Catheter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Central venous catheters are common in modern health care and are being increasingly used in both intensive care units and general wards. The primary aim of this study is to determine the incidence of mechanical complications within 24 hours after central venous catheterisation. The secondary aim is to identify risk factors associated with mechanical complications within 24 hours after catheterisation.

DETAILED DESCRIPTION:
Central venous catheters provide reliable access to the bloodstream, which allows delivery of medications and nutritional support that cannot be given safely through peripheral venous catheters.

Mechanical complications of central venous catheterisation include bleeding (such as hematoma and hemothorax), cardiac arrhythmia, arterial puncture, arterial catheterisation, nerve injury, pneumothorax, failed catheterisation and catheter tip malposition. The most common mechanical complications are arterial puncture, hematoma formation and pneumothorax. The number of mechanical complications related to central venous catheterisation varies widely in previous studies with incidences between 1.1 and 34 %. Ultrasound guidance reduces the incidence of mechanical complications, but despite evidence demonstrating improved safety, real-time ultrasound guidance is still not routinely used by all physicians when obtaining central venous access.

Four hospitals in Region Skåne, Sweden, will participate in this study: one university hospital with approximately 1300 beds and three county hospitals with about 200 beds each. All central venous catheter insertions at the participating hospitals during the study period will be included in the study.

The primary aim of this prospective, controlled, observational study is to determine the incidence of mechanical complications within 24 hours after central venous catheterisation. The secondary aim is to identify independent risk factors of mechanical complications within 24 hours after insertion of central venous catheters.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving a central venous catheter will be observed

Exclusion Criteria:

* Patients that dies within 24 hours after insertion of a central venous catheter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients at the included hospitals who are receiving a central venous catheter insertions during the study period will be observed
Sampling Method: Non-Probability Sample
Enrollment: 12600 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of cases with bleeding grade 3-4 | Up to 24 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Grade 3 bleedings/hematoma formation/hemothorax (bleedings requiring invasive intervention or blood transfusion) and grade 4 bleedings/hemothorax (life-threatening bleedings). Will be detected during the catheterisation or at the daily inspection by the patient responsible physician or nurse. Will be classified as major mechanical complications
Number of cases with bleeding grad 2 | Up to 24 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Grade 2 bleedings/hematoma formation (bleedings requiring external compression). Will be detected during the inserting procedure or at the daily inspection by the patient responsible physician or nurse. Will be considered minor mechanical complications.
Number of cases with pneumothorax at post-procedural x-ray of the thorax | Up to 24 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Pneumothoraces will be detected using x-ray after the central venous catheter insertion. All pneumothoraces will be classified as major mechanical complications
Number of cases with arterial puncture evident at the insertion procedure by the inserting physician | During the procedure of inserting the central venous catheter
  Mechanical complication after CVC-insertion. Will be detected by the inserting anesthesiologist and documented in the electronic chart. Will be considered a minor mechanical complication.
Number of cases with arterially positioned catheter at post-procedural x-ray | Up to 24 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Will be detected at a post-procedural x-ray of the thorax. Will be considered a major mechanical complication.
Number of cases with persistent nerve injury classified as sensory loss, paraesthesia or loss of motor neuron function recognized by the responsible physician or nurse | Persistent more than 72 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Will be detected and documented by the patient responsible physician or nurse. Will be considered a major mechanical complication.
Number of cases with transient nerve injury classified as sensory loss, paraesthesia or loss of motor neuron function recognized by the responsible physician or nurse | Transient up to 72 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Will be detected and documented by the patient responsible nurse. Will be considered a minor mechanical complication.
Number of cases with arrhythmia grad 3-4 during the inserting procedure | During the procedure of inserting the central venous catheter
  Mechanical complication during the CVC-insertion. Recognized at the continuous ECG by the inserting physician or the assistant. Arrhythmias grade 3 (symptomatic arrhythmia requiring urgent medical intervention) and grade 4 (symptomatic arrhythmia with life-threatening consequences) will be considered major mechanical complications.
Number of cases with arrhythmia grad 1-2 during the inserting procedure | During the procedure of inserting the central venous catheter
  Mechanical complication during the CVC-insertion. Recognized at the continuous ECG by the inserting physician or the assistant. Arrhythmias grade 1 (asymptomatic arrhythmia not requiring intervention) and grade 2 (asymptomatic or symptomatic arrhythmia requiring non-urgent medical intervention) will be considered minor mechanical complications.
Number of cases with failure to place the catheter | During the procedure of inserting the central venous catheter
  An attempt to insert a central venous catheter was performed but failed. Will be detected by the inserting anesthesiologist. Minor mechanical complications.
Number of cases with catheter tip malposition at post-procedural x-ray, where correction is needed before use | Up to 24 hours after insertion of central venous catheter
  Mechanical complication after CVC-insertion. Will be detected at a post-procedural x-ray of the thorax. Minor mechanical complications.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kander, Ass. Prof., Principal Investigator — Skane University Hospital
Locations (1):
- Region Skåne, Lund, Skåne County, Sweden

REFERENCES:
- [Derived] Naddi L, Hubinette J, Kander T, Borgquist O, Adrian M. Operator gender differences in major mechanical complications after central line insertions: a subgroup analysis of a prospective multicentre cohort study. BMC Anesthesiol. 2024 Feb 21;24(1):68. doi: 10.1186/s12871-024-02455-3. PMID 38383304
- [Derived] Adrian M, Borgquist O, Kroger T, Linne E, Bentzer P, Spangfors M, Akeson J, Holmstrom A, Linner R, Kander T. Mechanical complications after central venous catheterisation in the ultrasound-guided era: a prospective multicentre cohort study. Br J Anaesth. 2022 Dec;129(6):843-850. doi: 10.1016/j.bja.2022.08.036. Epub 2022 Oct 22. PMID 36280461
- [Derived] Adrian M, Borgquist O, Bentzer P, Akeson J, Spangfors M, Wrigstad J, Holmstrom A, Linner R, Kander T. Research protocol for mechanical complications after central venous catheterisation: a prospective controlled multicentre observational study to determine incidence and risk factors of mechanical complications within 24 hours after cannulation. BMJ Open. 2019 Oct 19;9(10):e029301. doi: 10.1136/bmjopen-2019-029301. PMID 31630102